CLINICAL TRIAL: NCT02945943
Title: Effects of a Six-week Rehabilitation Program in Conjunction With Thrust Mobilization on Lower Extremity Function in Subjects Reporting Chronic Ankle Instability
Brief Title: Effects of Mobilization in Conjunction With Therapeutic Exercise in Participants With a History of Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Cameron Jones, Assistant Professor Division of Physical Therapy, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-1627
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Functional Deficits; Manipulation; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Mobilization (Experimental): High Velocity Low Amplitude mobilization group. The three joints manipulated included proximal tibiofibular, the distal tibiofibular, and talocrural joints and were mobilized the first three sessions prior to the participants performing the exercise protocol.
  Interventions: Other: High Velocity Low Amplitude mobilization; Other: Exercise Protocol
- Exercise Protocol (Active Comparator): This exercise regimen is a modified version of the balance training program described by McKeon et al.
  Interventions: Other: Exercise Protocol

INTERVENTIONS:
Other: High Velocity Low Amplitude mobilization — Mobilizations were performed one time at each joint, prior to completing the exercise protocol during the first three treatment sessions.
  Other Names: HVLA; thrust mobilization
  Arms: Mobilization
Other: Exercise Protocol — This exercise regimen is a modified version of the balance training program described by McKeon et al.
  Other Names: Control

SUMMARY:
Our purpose was to examine the combined effects of thrust mobilization of the proximal and distal ankle joints in conjunction with a six-week rehabilitation program on ankle function in subjects reporting chronic ankle instability (CAI).

DETAILED DESCRIPTION:
Joint mobilizations are reported to increase range of motion (ROM), postural control and proprioception, and decrease pain in individuals with CAI. There is no research supporting the combined effects of thrust mobilization and exercise on function in this population.

Inclusion and exclusion criterion were established and a convenience sample was performed. 19 subjects were randomized into the exercise only or mobilization (experimental) and exercise group. Both groups underwent 12 supervised training sessions across a six-week period. The mobilization (experimental) group also received high-velocity-low-amplitude (HVLA) thrust mobilizations at the talocrural, proximal, and distal tibiofibular joints prior to the first three treatment sessions.

An examiner blinded to involved limb and group allocation performed a baseline and six-week follow-up examination of muscle strength, joint mobility, range of motion, and/or functional performance. The participants completed subjective outcome measures at baseline, 2 weeks, 4 weeks, and finally at 6 weeks including the Functional Ankle Disability Index (FADI), FADI-Sport, and the Ankle Joint Functional Assessment Tool (AJFAT). Participants also completed baseline and a six-week follow up assessments of the figure-of-8 hop test, side hop test, and three directions of the Star Excursion Balance test (SEBT).

The exercise protocol is a modified version of the balance training program described by McKeon et al. Participants completed this protocol twice a week, for six weeks. Treatment sessions lasted approximately 30 minutes. Participants were individually progressed on particular exercises if zero errors were observed. In addition, all participants were given a home exercise program (HEP) to complete every day of the week excluding treatment days.

The mobilization (experimental) group received HVLA thrust mobilizations at the three joints stated above for the first three sessions prior to completing the exercise protocol. Each mobilization was performed one time at each joint. The order of joint mobilizations was randomized prior to administering.

Data analysis was performed using International Business Machines Statistical Package for the Social Sciences (SPSS) version (22). Alpha level was set p<0.05. Separate 2 x 2 repeated measures analysis of variance (ANOVA) were used to assess changes in the FADI, FADI-Sport, figure-of-8 hop test, side hop test, and three directions of the SEBT.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 35 years old age
* Self-reported history of an ankle sprain
* Reports of "giving way" or a "loose" ankle within the past 6 months and/or decrease in functional status as compared to the uninvolved ankle

Exclusion Criteria:

* Lower extremity injury within the past 3 months
* History of vestibular dysfunction, neuromuscular diagnosis, mental illness, or if the participant was currently participating in another supervised rehabilitation program for the involved ankle.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline Figure-of-8 hop test at 6 weeks. | Baseline and 6 weeks
  The participant began the test on either side of a demarcated 5-meter distance. While standing on the involved ankle, the participant was instructed to "hop on one foot, as fast as you can," twice around the figure 8. Two trials were performed with the fastest time being recorded.
Change in baseline Side hop test at 6 weeks. | Baseline and 6 weeks
  The participant stands on the involved limb on either side of two lines that are 30 cm apart. They were then instructed to "hop on one foot, as fast as you can," laterally and then back to the starting position. This was counted as two repetitions and 10 repetitions were performed. If the participant landed on or between the lines, this repetition was not counted and they continued until 10 good repetitions were completed. Participants performed two trials and the fastest time was recorded.
Change in baseline Star Excursion Balance Test (SEBT) at 6 weeks. | Baseline and 6 weeks
  Each participant was asked to maintain single-limb stance, with hands on their hips, while reaching in anterior, posteromedial, and posterolateral directions.
Change in baseline Functional Ankle Disability Index (FADI) at 6 weeks. | Baseline, 2 week, 4 weeks, 6 weeks
  The FADI is a 26-item tool that is designed to assess functional limitations related to foot and ankle conditions. Each item is scored from 0 (unable to do) to 4 (no difficulty at all) and has total point value of 104 points.
Change in baseline Functional Ankle Disability Index (FADI)- Sport at 6 weeks. | Baseline, 2 week, 4 weeks, 6 weeks
  The FADI-Sport is an 8-item tool that is a sub-scale of the FADI. Each item is scored with from 0 (unable to do) to 4 with a total point value of 32 points, reported as a percent value.
Change in baseline Ankle Joint Functional Assessment Tool (AJFAT) at 6 weeks. | Baseline, 2 week, 4 weeks, 6 weeks
  12-item tool that rates the participant's overall perceived level of function. Each item is assigned a point value from 0 (much less than other ankle) to 4 (much more than other ankle) with a possible total value of 48 points.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R Jones, DPT, Principal Investigator — Shenandoah University Division of Physical Therapy; Sheri Hale, PhD, PT, Principal Investigator — Shenandoah University Division of Physical Therapy
Locations (1):
- Shenandoah University Division of Physical Therapy, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from subjective and objective outcome measures from all participants obtained prior to and after intervention have been analyzed.

REFERENCES:
- [Background] McKeon PO, Ingersoll CD, Kerrigan DC, Saliba E, Bennett BC, Hertel J. Balance training improves function and postural control in those with chronic ankle instability. Med Sci Sports Exerc. 2008 Oct;40(10):1810-9. doi: 10.1249/MSS.0b013e31817e0f92. PMID 18799992
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Hertel J. Sensorimotor deficits with ankle sprains and chronic ankle instability. Clin Sports Med. 2008 Jul;27(3):353-70, vii. doi: 10.1016/j.csm.2008.03.006. PMID 18503872
- [Background] Wikstrom EA, Hubbard TJ. Talar positional fault in persons with chronic ankle instability. Arch Phys Med Rehabil. 2010 Aug;91(8):1267-71. doi: 10.1016/j.apmr.2010.04.022. PMID 20684909
- [Background] Hale SA, Hertel J, Olmsted-Kramer LC. The effect of a 4-week comprehensive rehabilitation program on postural control and lower extremity function in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2007 Jun;37(6):303-11. doi: 10.2519/jospt.2007.2322. PMID 17612356
- [Background] Hupperets MD, Verhagen EA, van Mechelen W. Effect of unsupervised home based proprioceptive training on recurrences of ankle sprain: randomised controlled trial. BMJ. 2009 Jul 9;339:b2684. doi: 10.1136/bmj.b2684. PMID 19589822
- [Background] Beazell JR, Grindstaff TL, Sauer LD, Magrum EM, Ingersoll CD, Hertel J. Effects of a proximal or distal tibiofibular joint manipulation on ankle range of motion and functional outcomes in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2012 Feb;42(2):125-34. doi: 10.2519/jospt.2012.3729. Epub 2012 Feb 1. PMID 22333567
- [Background] Hubbard TJ, Hertel J. Anterior positional fault of the fibula after sub-acute lateral ankle sprains. Man Ther. 2008 Feb;13(1):63-7. doi: 10.1016/j.math.2006.09.008. Epub 2006 Dec 26. PMID 17188923
- [Background] Denegar CR, Hertel J, Fonseca J. The effect of lateral ankle sprain on dorsiflexion range of motion, posterior talar glide, and joint laxity. J Orthop Sports Phys Ther. 2002 Apr;32(4):166-73. doi: 10.2519/jospt.2002.32.4.166. PMID 11949665
- [Background] Grindstaff TL, Beazell JR, Sauer LD, Magrum EM, Ingersoll CD, Hertel J. Immediate effects of a tibiofibular joint manipulation on lower extremity H-reflex measurements in individuals with chronic ankle instability. J Electromyogr Kinesiol. 2011 Aug;21(4):652-8. doi: 10.1016/j.jelekin.2011.03.011. Epub 2011 May 4. PMID 21546263
- [Background] Whitman JM, Childs JD, Walker V. The use of manipulation in a patient with an ankle sprain injury not responding to conventional management: a case report. Man Ther. 2005 Aug;10(3):224-31. doi: 10.1016/j.math.2004.10.003. Epub 2005 Jan 21. No abstract available. PMID 16038858
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342